CLINICAL TRIAL: NCT06976502
Title: Health eHeart BioBank
Acronym: HeH BioBank
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 24-40979
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Heart Diseases; Cardiac Diseases; Vascular Diseases; Cardiovascular Diseases
Keywords: Heart Disease; Cardiovascular Disease; Cardiology
MeSH Terms: conditions — Heart Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood samples with be collected with the option of DNA, heart tissue, and other samples may be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with a History of Cardiovascular Disease
  Interventions: Procedure: Blood Draw; Procedure: Tissue Collection; Procedure: DNA Collection; Other: Medical Chart Review
- Participants with a Family History of Cardiovascular Disease
  Interventions: Procedure: Blood Draw; Procedure: Tissue Collection; Procedure: DNA Collection; Other: Medical Chart Review
- Healthy Controls
  Interventions: Procedure: Blood Draw; Procedure: Tissue Collection; Procedure: DNA Collection; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Blood Draw — Participants will be asked to contribute approximately 36 mL of blood using standard procedures and obtained at the time of a clinically ordered routine blood draw or a study ordered blood draw. Participants may be asked to contribute additional blood samples over the course of their participation in the study.
Procedure: Tissue Collection — If the participant is undergoing a clinically ordered procedure (e.g. heart surgery/biopsy/transplant), then they will be asked to contribute tissue to the study before any tissue is collected during the procedure. Most samples collected by the HeH BioBank will be tissue that would be normally discarded after the procedure.
Procedure: DNA Collection — Participants will be asked to contribute their DNA for Whole Genome Sequencing (WGS) to help identify genetic markers of heart disease. DNA will be obtained at the time of the blood draw or obtained through DNA collection kits administered to participants who are unable or unwilling to undergo a blood draw.
Other: Medical Chart Review — Demographic, clinical, and pathologic information will be extracted from the participant's medical record.
  Other Names: Medical Record Review

SUMMARY:
The purpose of the Health eHeart BioBank is to collect and store specimen (e.g. blood, DNA, tissue) for future studies at the University of California, San Francisco (UCSF) that will help determine changes and identify molecular and genetic markers in the human body that might help increase our knowledge of heart disease and guide development of new diagnostic tools and treatments that may help rapidly detect heart disease and prevent and/or treat heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older.

And at least one of the following:

* Established patient seen at UCSF and/or is a current participant in a clinical study that utilizes the HeH BioBank for biospecimen collection.
* Family member of a patient with cardiovascular disease.
* Patient with no cardiovascular disease.

Exclusion Criteria:

* Unwilling to consent to biospecimen collection through the HeH BioBank.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population are patients of the University of California, San Francisco and their relatives.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Establish and Maintain a Centralized Biorepository | Up to 10 years
  Establish and maintain a centralized biorepository to collect and store a variety of biospecimen samples and clinical data.
  This would allow for the samples and clinical data to be used to test hypotheses regarding the molecular and genetic basis of diagnosis and treatment of cardiovascular diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Olgin, MD, Principal Investigator — University of California, San Francisco; Gregory Marcus, MD, Principal Investigator — University of California, San Francisco; Vasanth Vedantham, MD, Principal Investigator — University of California, San Francisco; Connor G O'Brien, MD, Principal Investigator — University of California, San Francisco; James P Pirruccello, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rahmutula D, Marcus GM, Wilson EE, Ding CH, Xiao Y, Paquet AC, Barbeau R, Barczak AJ, Erle DJ, Olgin JE. Molecular basis of selective atrial fibrosis due to overexpression of transforming growth factor-beta1. Cardiovasc Res. 2013 Sep 1;99(4):769-79. doi: 10.1093/cvr/cvt074. Epub 2013 Apr 23. PMID 23612580
- [Background] Tseng ZH, Olgin JE, Vittinghoff E, Ursell PC, Kim AS, Sporer K, Yeh C, Colburn B, Clark NM, Khan R, Hart AP, Moffatt E. Prospective Countywide Surveillance and Autopsy Characterization of Sudden Cardiac Death: POST SCD Study. Circulation. 2018 Jun 19;137(25):2689-2700. doi: 10.1161/CIRCULATIONAHA.117.033427. PMID 29915095
- [Background] Aouizerat BE, Vittinghoff E, Musone SL, Pawlikowska L, Kwok PY, Olgin JE, Tseng ZH. GWAS for discovery and replication of genetic loci associated with sudden cardiac arrest in patients with coronary artery disease. BMC Cardiovasc Disord. 2011 Jun 10;11:29. doi: 10.1186/1471-2261-11-29. PMID 21658281
- [Background] Roberts JD, Hsu JC, Aouizerat BE, Pullinger CR, Malloy MJ, Kane JP, Olgin JE, Marcus GM. Impact of a 4q25 genetic variant in atrial flutter and on the risk of atrial fibrillation after cavotricuspid isthmus ablation. J Cardiovasc Electrophysiol. 2014 Mar;25(3):271-277. doi: 10.1111/jce.12317. Epub 2013 Dec 13. PMID 24237655
- [Background] Roberts JD, Dewland TA, Glidden DV, Hoffmann TJ, Arking DE, Chen LY, Psaty BM, Olgin JE, Alonso A, Heckbert SR, Marcus GM. Impact of genetic variants on the upstream efficacy of renin-angiotensin system inhibitors for the prevention of atrial fibrillation. Am Heart J. 2016 May;175:9-17. doi: 10.1016/j.ahj.2016.02.002. Epub 2016 Feb 13. PMID 27179719
- [Background] Roberts JD, Dewland TA, Longoria J, Fitzpatrick AL, Ziv E, Hu D, Lin J, Glidden DV, Psaty BM, Burchard EG, Blackburn EH, Olgin JE, Heckbert SR, Marcus GM. Telomere length and the risk of atrial fibrillation: insights into the role of biological versus chronological aging. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1026-32. doi: 10.1161/CIRCEP.114.001781. Epub 2014 Nov 8. PMID 25381796
- [Background] Marcus GM, Smith LM, Glidden DV, Wilson E, McCabe JM, Whiteman D, Tseng ZH, Badhwar N, Lee BK, Lee RJ, Scheinman MM, Olgin JE. Markers of inflammation before and after curative ablation of atrial flutter. Heart Rhythm. 2008 Feb;5(2):215-21. doi: 10.1016/j.hrthm.2007.10.007. Epub 2007 Oct 7. PMID 18242542
- [Background] Roberts JD, Longoria J, Poon A, Gollob MH, Dewland TA, Kwok PY, Olgin JE, Deo RC, Marcus GM. Targeted deep sequencing reveals no definitive evidence for somatic mosaicism in atrial fibrillation. Circ Cardiovasc Genet. 2015 Feb;8(1):50-7. doi: 10.1161/CIRCGENETICS.114.000650. Epub 2014 Nov 18. PMID 25406240
- [Background] Marcus GM, Rosenthal DG, Nah G, Vittinghoff E, Fang C, Ogomori K, Joyce S, Yilmaz D, Yang V, Kessedjian T, Wilson E, Yang M, Chang K, Wall G, Olgin JE. Acute Effects of Coffee Consumption on Health among Ambulatory Adults. N Engl J Med. 2023 Mar 23;388(12):1092-1100. doi: 10.1056/NEJMoa2204737. PMID 36947466